CLINICAL TRIAL: NCT06518928
Title: SprmPik AI Assisted Sperm Selection Study, an Assistant for Sperm Selection During ICSI
Brief Title: SprmPik AI Sperm Selection Study SiD, an Assistant for Sperm Selection During Intracytoplasmic Sperm Injection in Medically Assisted Reproduction: Effect on Fertilization, Blastocyst Formation, Early Pregnancy Loss, and Consistent Practice. A Prospective Pilot Study.
Acronym: SprmPik
Status: Recruiting | Type: Observational
Sponsor: Ovation Fertility (Other)
Collaborators: IVF 2.0 Limited (Other)
Responsible Party: Sponsor
Other Study IDs: OVA-9-2022-TX
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AI Asssited Sperm Selection: SiD software to select sperm for ICSI
  Interventions: Other: Artificial Intelligence assisted sperm selection
- Manual Sperm Selection: Human visualization of sperm for ICSI selection

INTERVENTIONS:
Other: Artificial Intelligence assisted sperm selection — SiD software for sperm selection
  Groups: AI Asssited Sperm Selection

SUMMARY:
SprmPik AI Assisted Sperm Selection Study SiD, an assistant for sperm selection during intracytoplasmic sperm injection in medically assisted reproduction: effect on fertilization, blastocyst formation, early pregnancy loss, and consistent practice. A prospective pilot study.

DETAILED DESCRIPTION:
The purpose of this research is to evaluate the impact of sperm selection for ICSI using the investigational SiD software, on performance outcomes such as the rate of fertilization, blastocyst development, clinical pregnancy success, and other intermediate results, in a pilot study.

SiD is a software designed to identify, evaluate, and assist in the sperm selection process within a semen sample, according to motility (for instance velocity, linearity, straightness) patterns and the shape of the sperm. SID uses a mathematical model. Its purpose is to assist clinical embryologists in selecting sperm to inject during ICSI. Currently, embryologists identify and select sperm based on the sperm motility and shape; not using any mathematical interphase assistant.

ELIGIBILITY:
Inclusion criteria for Male Partner (sperm source)

* Informed consent signed by the patient before treatment.
* IVF treatments with medical or embryology indication to perform ICSI.
* Fresh or frozen ejaculated motile sperm.
* Selection of sperm using a 7% or 10% PVP solution.
* Presence of motile sperm at the time of sperm selection for ICSI.
* Partner sperm

Exclusion criteria for Male Partner (sperm source)

* Sperm extracted by testicular biopsy.
* That the recommendations for use of SiD have not been fully followed.
* Inability to reliably trace sperm-oocyte-embryo throughout the process.
* Patients with immotile sperm

Inclusion criteria for Female Partner (egg source)

* Informed consent signed by the patient before treatment.
* IVF treatments with medical or embryology indication to perform ICSI.
* Cycles with at least 4 mature oocytes (Metaphase II).
* Fresh or frozen oocytes.

Exclusion criteria for Female Partner (egg source)

* Inability to reliably trace sperm-oocyte-embryo throughout the process.
* Oocytes that are not in Metaphase II.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients seeking fertility treatment by ICSI.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Oocyte Fertilization | 1 day
  Does SiD assist in ICSI Fertilization

SECONDARY OUTCOMES:
Blastocyst Formation | 7 days
  Do embryos develop better from SiD oocytes

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Ovation Fertility Las Vegas, Las Vegas, Nevada
  - Ovation Fertility - Austin, Austin, Texas